CLINICAL TRIAL: NCT02914561
Title: Combined Phase 3, Double-blind, Randomized, Placebo-Controlled Studies Evaluating the Efficacy and Safety of Filgotinib in the Induction and Maintenance of Remission in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Filgotinib in the Induction and Maintenance of Remission in Adults With Moderately to Severely Active Crohn's Disease
Acronym: DIVERSITY1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-419-3895; 2016-001367-36 (EudraCT Number)
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort A: Filgotinib 200 (mg) (Induction Study) (Experimental): Biologic naïve and biologic experienced participants received filgotinib 200 milligram (mg) with placebo-to-match (PTM) filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Cohort A: Filgotinib 100 mg (Induction Study) (Experimental): Biologic naïve and biologic experienced participants received filgotinib 100 mg with PTM filgotinib 200 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Cohort A: Placebo (Induction Study) (Placebo Comparator): Biologic naïve and biologic experienced participants received PTM filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Cohort B: Filgotinib 200 mg (Induction Study) (Experimental): Biologic experienced participants received filgotinib 200 mg with PTM filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Cohort B: Filgotinib 100 mg (Induction Study) (Experimental): Biologic experienced participants received filgotinib 100 mg with PTM filgotinib 200 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Cohort B: Placebo (Induction Study) (Placebo Comparator): Biologic experienced participants received PTM filgotinib 200 mg with PTM filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
  Interventions: Drug: Filgotinib; Other: Placebo
- Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) (Experimental): Participants who received filgotinib 200 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, up to Week 58.
  Interventions: Drug: Filgotinib
- Filgotinib 200 mg to Placebo (Maintenance Study) (Experimental): Participants who received filgotinib 200 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
  Interventions: Drug: Filgotinib; Other: Placebo
- Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) (Experimental): Participants who received filgotinib 100 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received filgotinib 100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
  Interventions: Drug: Filgotinib
- Filgotinib 100 mg to Placebo (Maintenance Study) (Experimental): Participants who received filgotinib 100 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, up to Week 58.
  Interventions: Drug: Filgotinib; Other: Placebo
- Placebo to Placebo (Maintenance Study) (Placebo Comparator): Participants who received placebo in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Filgotinib — Filgotinib tablets administered orally once daily.
  Other Names: GS-6034; GLPG0634
  Arms: Cohort A: Filgotinib 100 mg (Induction Study); Cohort A: Filgotinib 200 (mg) (Induction Study); Cohort A: Placebo (Induction Study); Cohort B: Filgotinib 100 mg (Induction Study); Cohort B: Filgotinib 200 mg (Induction Study); Cohort B: Placebo (Induction Study); Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study); Filgotinib 100 mg to Placebo (Maintenance Study); Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study); Filgotinib 200 mg to Placebo (Maintenance Study)
Other: Placebo — Placebo administered orally once daily.
  Arms: Cohort A: Filgotinib 100 mg (Induction Study); Cohort A: Filgotinib 200 (mg) (Induction Study); Cohort A: Placebo (Induction Study); Cohort B: Filgotinib 100 mg (Induction Study); Cohort B: Filgotinib 200 mg (Induction Study); Cohort B: Placebo (Induction Study); Filgotinib 100 mg to Placebo (Maintenance Study); Filgotinib 200 mg to Placebo (Maintenance Study); Placebo to Placebo (Maintenance Study)

SUMMARY:
The primary objectives of this study are to evaluate the safety and efficacy of filgotinib during induction and maintenance treatment of moderately to severely active Crohn's disease (CD) in participants who are biologic-naive and biologic-experienced.

Participants who complete the study, or do not meet protocol response or remission criteria at Week 10 will have the option to enter a separate long-term extension (LTE) study (Study GS-US-419-3896).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of CD with a minimum disease duration of 3 months with involvement of the ileum and/or colon at a minimum, as determined by histopathology and endoscopic assessment
* Moderately to severely active CD
* Cohort A (Biologic Naïve): Previously demonstrated an inadequate clinical response, loss of response to, or intolerance to at least 1 of the following agents (depending on current country treatment recommendations/guidelines): corticosteroids and immunomodulators
* Cohort A (Biologic Experienced): Previously demonstrated an inadequate clinical response, loss of response to, or intolerance to at least 1 of the following agents (depending on current country treatment recommendations/guidelines) or discontinuation of use of at least one of the following agents for reasons other than inadequate clinical response, loss of response or intolerance: tumor necrosis factor alpha (TNFa) antagonists, vedolizumab, and ustekinumab
* Cohort B (Biologic Experienced): Previously demonstrated an inadequate clinical response, loss of response to, or intolerance to at least 1 of the following agents (depending on current country treatment recommendations/guidelines): TNFa antagonists, vedolizumab, and ustekinumab

Key Exclusion Criteria:

* Current complications of CD such as symptomatic strictures, severe rectal/anal stenosis, fistulae other than perianal fistulae, short bowel syndrome, etc.
* Presence of ulcerative colitis, indeterminate colitis, ischemic colitis, fulminant colitis, or toxic mega-colon
* Active tuberculosis (TB) or history of latent TB that has not been treated
* Use of any prohibited concomitant medications as described in the study protocol

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1372 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (513):
- United States (101):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Southern California Research Center, Inc., Coronado, California
  - VVCRD Research, Garden Grove, California
  - UC San Diego Health System, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Inland Empire Clinical Trials, LLC, Rialto, California
  - Kaiser Permanente, San Francisco, California
  - Clearview Medical Research, LLC, Santa Clarita, California
  - University of Colorado Denver and Hospital, Aurora, Colorado
  - South Denver Gastroenterology, PC, Lone Tree, Colorado
  - Connecticut GI, PC-Research Division, Farmington, Connecticut
  - Medstar Georgetown University Hospital (Patient Exams), Washington D.C., District of Columbia
  - Advanced Research, LLC, Coral Springs, Florida
  - UF Clinical Research Center, Gainesville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Florida Center for Gastroenterology, Largo, Florida
  - University of Miami Crohn's and Colitis Center, Miami, Florida
  - Advanced Pharma CR, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Vista Health Research, LLC, Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Center for Interventional Endoscopy - AdventHealth Orlando, Orlando, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Tampa General Hospital, Tampa, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Atlanta Gastroenterology Specialist, PC, Suwanee, Georgia
  - Illinois Gastroenterology Group - Arlington Heights, Arlington Heights, Illinois
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Illinois Gastroenterology Group - Gurnee, Gurnee, Illinois
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, School of Medicine, Louisville, Kentucky
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Investigative Clinical Research, Annapolis, Maryland
  - University of Maryland Medical Center, Baltimore, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Massachusetts General Hospital - Crohn's and Colitis Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Spectrum Health Butterworth Hospital, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - NY Scientific, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - New York University School of Medicine/NYU Gastroenterology Associates, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Charlotte Gastroenterology & Hepatology, PLLC, Charlotte, North Carolina
  - Carolina's GI Research, LLC, Raleigh, North Carolina
  - Fargo Gastroenterology and Hepatology Clinic, Fargo, North Dakota
  - Consultants for Clinical Research, Cincinnati, Ohio
  - UC Health Physicians Clifton, Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC,, Mentor, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - Options Health Research LLC, Tulsa, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Vanderbilt University Medical Center - IBD Clinic, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - DHAT Research Institute, Garland, Texas
  - Kelsey-Seybold Clinic, Houston, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Gulf Coast Research Group, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - TDDC San Marcos, San Marcos, Texas
  - Texas Digestive Disease Consultants (IP Shipment), Southlake, Texas
  - Spring Gastroenterology, The Woodlands, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - HP Clinical Research, Bountiful, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Emeritas Research Group LLC, Leesburg, Virginia
  - McGuire DVAMC, GI (111N), Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, a division of GI Associates, LLC, Milwaukee, Wisconsin
- Fundacion Estudios Clinicos CiRec, Rosario, Argentina
- Australia (17):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, New South Wales
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Coastal Digestive Health, Mountain Creek, Queensland
  - Coral Sea Clinical Research Institute (Mackay), North Mackay, Queensland
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Emeritus Research, Camberwell, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Universitatsklinik Innsbruck, Innsbruck
  - AKH-Medizinische Universitat Wien, Vienna
- Belgium (8):
  - GZA Ziekenhuizen campus Sint-Vincentius, Antwerp
  - Imelda General Hospital, Bonheiden
  - CUB Hopital Erasme, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Chretien (CHC) - Clinique Saint-Joseph, Liège
  - CHR Citadelle, Liège
  - AZ Delta Campus Wilgenstraat, Roeselare
- Bulgaria (4):
  - Medical Center - Complete Medical Solutions OOD, Samokov
  - Medical Center - "Tsaritsa Yoanna" EOOD, Sliven
  - "MDHAT Dr. St.Cherkezov" AD, Veliko Tarnovo
  - MHAT "Sveta Petka" AD, Vidin
- Canada (10):
  - Barrie GI Associates, Barrie
  - University of Calgary, Heritage Medical Research Clinic, Calgary
  - Hamilton Health Sciences Corporation, McMaster University Medical Centre, Hamilton
  - London Health Sciences Centre - University Hospital, London
  - TIDHI Innovation Inc., North York
  - ABP Research Services, Oakville
  - Royal University Hospital, Saskatoon
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver
  - Toronto Digestive Disease Associates Inc., Vaughan
  - Percuro Clinical Research Ltd., Victoria
- Croatia (3):
  - University Hospital Center Osijek, Osijek
  - Clinical Hospital Dubrava, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (5):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Oblastni nemocnice Mlada Boleslav, a.s., nemocnice Stredoceskeho kraje, Gastroenterologicke oddeleni, Mladá Boleslav
  - G.E.P. Clinic, s r.o., Prague
  - Thomayerova nemocnice, Interni klinika 3. LF UK a TN (Interni Oddeleni), Prague
  - ISCARE a.s. (Klinicke centrum ISCARE), Klinicke a vyzkumne centrum pro strevni zanety, Prague
- France (23):
  - CHU Amiens Picardie, Amiens
  - CHU de Caen, Caen
  - CHU de Clermont-Ferrand - Hopital d'Estaing, Clermont-Ferrand
  - APHP - Hopital Beaujon - Clichy - Universite Paris VII, Clichy
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - CHU de Dijon Bourgogne - Hopital Francois Mitterand, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Hopital Universitaire de Bicetre, Le Kremlin-Bicêtre
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hopital Nord, Marseille
  - Hopital Saint Joseph, Marseille
  - CHU de Montpellier-Hopital Saint Eloi, Montpellier
  - Centre d'Investigation Clinique - CHU Hotel-Dieu, Nantes
  - Hopital de l'Archet 2, Nice
  - CHU de Bordeaux - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire de Lyon Sud, Pierre-Bénite
  - CH Annecy Genevois - Site d'Annecy, Pringy
  - Centre Hospitalier Universitaire de Rennes - Hopital Pontchaillou, Rennes
  - CHU de Saint-Etienne - Hopital Nord, Saint-Priest-en-Jarez
  - Nouvel Hopital Civil, Strasbourg
  - Hopitaux Universitaires de Strasbourg - Hopital de Hautepierre, Strasbourg
  - CHU de Toulouse - Hopital Rangueil, Toulouse
  - CHU de Nancy - Hopital Brabois Adultes, Vandœuvre-lès-Nancy
- Georgia (3):
  - Unimed Ajara LLC - Batumi Referral Hospital, Batumi
  - Medi Club Georgia LLC, Tbilisi
  - Ltd. Unimed Kakheti - Telavi Referral Hospital, Telavi
- Germany (24):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Gastro-Studien, Berlin
  - Charite - Universitatsmedizin Berlin, Berlin
  - DRK Kliniken Berlin - Westend - Klinik fuer Innere Medizin, Berlin
  - Stadtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Universitatsklinik Koln, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - CED Studien UG, Interdisciplinary Crohn Colitis Center (iCCC) Rhein-Main, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Westklinikum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Heidelberg, Heidelberg
  - Praxis fur Gastroenterologie, Heidelberg
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Universitatsklinikum Jena, Jena
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - EUGASTRO GmbH, Leipzig
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Luneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitat Munchen - Grosshadern, München
  - Universitaetsmedizin Rostock, Zentrum fuer Innere Medizin, Rostock
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitatsklinikum Ulm, Zentrum Fur Innere Medizin, Ulm
- Greece (5):
  - General Hospital of Athens "Hippokratio", 2nd Internal Medicine Clinic of Athens University, Hepato-gastroenterology Unit, Athens
  - University General Hospital "Attikon", 2nd Propaedeutic Internal Medicine Dept. and Research Unit, Hepatogastroenterology Unit, Athens
  - University General Hospital of Ioannina, Gastroenterology Department, Internal Medicine Division, Ioannina
  - University General Hospital of Patras "Panagia I Voithia", Gastroenterology Department, Internal Medicine Division, Pátrai
  - General Hospital of Thessaloniki "Hippokratio", 4th Internal Medicine Department of Aristotle University of Thessaloniki, Thessaloniki
- Hong Kong (4):
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Department of Medicine & Therapeutics, The Chinese University of Hong Kong, Prince of Wales Hospital, Shatin
  - Tuen Mun Hospital, Tuenmen
- Hungary (8):
  - Bekes Megyei Kosponti Korhaz, Dr. Rethy Pal Tagkorhaz, IV. Belgyogyaszat - 2. Gasztroenterologia, Békéscsaba
  - Szent Margit Korhaz, Gasztroenterológiai Osztály, Budapest
  - Clinexpert Egeszsegugyi Szolgaltato es Kereskedelmi Kft., Budapest
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Kozponti Felnott Szakrendelo, Budapest
  - Szent Janos Korhaz es Eszak-budai Egitett Korhazak, I. Belgyogyaszati - Gasztroenterologiai Osztaly, Budapest
  - Debreceni Egyetem Klinikai Kozpont, II. sz. Belgyogyaszati Klinika, Gasztroenterologia, Debrecen
  - Bugat Pal Korhaz, Belgyogyaszat, Gyöngyös
  - Karolina Korhaz es Rendelointezet, Altalanos Belgyogyaszat-Gasztroenterologia, Mosonmagyaróvár
- Landspitali University Hospital, Reykjavik, Iceland
- India (50):
  - S.P. Medical College & AG of Hospitals, Bikaner, Rajasthan
  - Kaizen Hospital, Ahmedabad
  - Gastroplus Digestive Disease Centre Pvt Ltd, Ahmedabad
  - Sal Hospital and Medical Institute, Ahmedabad
  - Victoria Hospital, Bangalore Medical College and Research Institute, Bangalore
  - M S Ramaiah Medical College and Hospital, Bangalore
  - KLES Dr. Prabhakar Kore Hospital & MRC, Belagavi
  - BGS Global Hospital, Bengaluru
  - Apollo Speciality Hospital, Chennai
  - VGM Hospital Institute of Gastroenterology, Coimbatore
  - Maharaja Agrasen Hospital, Delhi
  - Lourdes Hospital, Ernākulam
  - PVS Memorial Hospital Private Limited, Ernākulam
  - Institute of Digestive & Liver Diseases, Guwahati
  - Fortis Medical Research Institute, Gūrgaon
  - Gleneagles Global Hospitals, Hyderabad
  - Citizens Specialty Hospital, Hyderabad
  - Aware Gleneagles Global Hospitals, Hyderabad
  - Centre for Liver Research & Diagnostics, Hyderabad
  - Asian Institute of Gastroenterology Pvt Ltd, Hyderabad
  - S.R.Kalla Memorial Gastro.&General Hospital, Jaipur
  - S.M.S Medical College & Hospitals, Jaipur
  - GSVM Medical College, Kanpur
  - Lakeshore Hospital and Research Centre Ltd., Kochi
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - School of Digestive & Liver Diseases, Kolkata
  - Apollo Gleneagles Hospitals, Kolkata
  - King George's Medical University, Lucknow
  - Dayanand Medical College & Hospital, Ludhiana
  - Kasturba Medical College (KMC) Hospital, Mangaluru
  - Seth G.S Medical College & KEM Hospital, Mumbai
  - Lokmanya Tilak Municipal General Hospital, Mumbai
  - Midas Multispeciality Hospital Pvt. Ltd, Nagpur
  - Suretech Hospital & Research Centre Ltd, Nagpur
  - Max Smart Super Speciality Hospital, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Dr. B.L. Kapur Memorial Hospital, New Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi
  - S.L Raheja Hospital, Pārel
  - Department of Surgery, B.J. Government Medical College & Sassoon General Hospital, Pune
  - Grant Medical Foundation Ruby Hall Clinic, Pune
  - Universal Hospital, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Gandhi Hospital, Secunderabad
  - Institute of Gastroenterology & Liver Disease. Sunshine Hospitals, Secunderabad
  - Surat Institute of Digestive Sciences, Surat
  - BAPS Pramukh Swami Hospital, Surat
  - Kasturba Hospital Medical College, Udupi
  - Sterling Hospital, Vadodara
  - Samvedna Hospital, Varanasi
- Ireland (4):
  - St. Vincent's University Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Wellcome Trust HRB Clinical Research Facility, Dublin
  - University Hospital Galway, Galway
- Israel (11):
  - Emek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kefar Sava
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - UOC Gastroenterologia II, Castellana Grotte
  - U.O. Fisiopatologia Digestiva, Catanzaro
  - UOC Medicina Interna, Cento
  - Ospedale Clinicizzato SS. Annunziata - Dipartimento di Medicina, Chieti
  - Gastroenterologia clinica - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Endoscopia Digestiva Centralizzata, Milan
  - UO Gastroenterologia, Modena
  - UOC Gastroenterologia, Padua
  - Azienda Ospedaliero-Universitaria Pisana - Presidio Ospedaliero Cisanello, Pisa
  - UOC di Gastroenterologia ed Endoscopia Digestiva, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O. Ordine Mauriziano di Torino, Torino
- Japan (49):
  - Ohmori Toshihide gastro-intestinal Clinic, Ageo-shi
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital, Chūōku
  - Japanese Red Cross Fukuoka Hospital, Fukuoka
  - Tokai University Hachioji Hospital, Hachiōji
  - Medical corporation Ryowakai, Hamamatsu South Hospital, Hamamatsu
  - Hiroshima Prefectural Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Fukuoka University Hospital, Jonan-ku
  - Nanpuh Hospital, Kagoshima
  - Ofuna Chuo Hospital, Kamakura
  - Tsujinaka Hospital, Kashiwa
  - Saitama Medical Center, Saitama Medical University, Kawagoe
  - Kitakyushu City Hospital Organization Kitakyushu Municipal Medical Center, Kitakyushu-shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Kurume University Hospital, Kurume-shi
  - Hidaka Coloproctology Clinic, Kurume-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - The Jikei University Hospital, Minatoku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka-shi
  - Iwate Medical University Hospital, Morioka
  - Aichi Medical University Hospital, Nagakute-shi
  - Nagasaki University Hospital, Nagasaki
  - Nagoya City University Hospital, Nagoya
  - Saiseikai Niigata Daini Hospital, Nishiku
  - Hyogo College of Medicine College Hospital, Nishinomiya
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - Osaka City University Hospital, Osaka
  - Wakakusa-Daiichi Hospital, Osaka
  - Ishida IBD Clinic, Ōita
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga-Ken Medical Centre Koseikan, Saga
  - Saga University Hospital, Saga
  - Kitasato University Hospital, THE KITASATO INSTITUTE, Sagamihara
  - Tokito Clinic, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - National Hospital Organization Sendai Medical Center, Sendai
  - Tokyo Yamate Medical Center, Shinjuku-ku
  - Osaka University Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki-shi
  - Osaka Medical College Hospital, Takatsuki
  - Ieda Hospital, Toyota-shi
  - Wakayama Medical University Hospital, Wakayama
  - Yokohama Health Medicine Association Kannai Suzuki Clinic, Yokohama
- Malaysia (5):
  - Universiti Kebangsaan Malaysia Medical Center, Cheras
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
- Netherlands (9):
  - NZW Alkmaar (Noordwest Ziekenhuisgroep), Alkmaar
  - VU University Medical Centre, Amsterdam
  - Academic Medical Center (AMC), Amsterdam
  - Gelre Hospital, Apeldoorn
  - University Medical Center Groningen (UMCG), Groningen
  - Maastricht University Medical Centre, Maastricht
  - Erasmus University Medical Center, Rotterdam
  - Elisabeth-TweeSteden Hospital, Tilburg
  - University Medical Center Utrecht, Utrecht
- New Zealand (7):
  - Christchurch Hospital, Christchurch
  - Southern District Health Board - Dunedin Hospital, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Newtown
  - Bay of Plenty District Health Board - Tauranga Hospital, Tauranga
  - Hutt Valley District Health Board - Hutt Valley Hospital, Wellington
- Vestre Viken Hospital Trust, Baerum Hospital, Drammen, Norway
- Poland (26):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Klinika Gastroenterologii i Chorob Wewnetrznych, Bialystok
  - VITAMED Galaj i Cichomski spolka jawna, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im. Dr. Jana Biziela w Bydgoszczy, Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych, Bydgoszcz
  - Gabinet Lekarski Janusz Rudzinski, Bydgoszcz
  - NZOZ INTER-MED, Centrum Endoskopowe, Częstochowa
  - Niepubliczny Zaklad Opieki Zdrowotnej ALL-MEDICUS, Katowice
  - Centrum Medyczno-Diagnostyczne Prima-Med, Krakow
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Uniwerstyeckiego Szpitala Klinicznego nr 1 im. Norbert Barlickiego, Lodz
  - Trialmed Crs, Piotrkow Trybunalski
  - Clinical Research Center Spolka z ograniczna odpowiedzialnoscia Medic-R Sp. k., Poznan
  - Gabinet Lekarski Dr. Hab. N. Med. Bartosz Korczowski, Rzeszów
  - Endoskopia Sp. Z o.o., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - GASTROMED Kopon, Zmudzkinski i Wspolnicy Sp. j. Specjalistyczne Centrum Gastrologii i Endoskopii, Torun
  - H-T.Centrum Medyczne Spolka z Ograniczona Odpowiedzialnoscia Sp.K., Tychy
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnetrznych i Administacji w Warszawie, Warsaw
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Medical Concierge Centrum Medyczne, Warsaw
  - Niepubliczny Zaklad Opieki Zrodotnej VIVAMED Jadwige Miecz, Warsaw
  - Bodyclinic, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Centrum Medyczne, Wroclaw
- Portugal (8):
  - Hospital de Braga, Braga
  - Centro Hospitalar e Universitario de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar Cova de Beira, EPE, Covilha
  - Centro Hospitalar do Algarve EPE, Faro
  - Hospital da Senhora da Oliveira Guimaraes, E.P.E., Guimarães
  - Hospital Beatriz Angelo, Loures
  - Centro Hospitalar de Sao Joao, EPE, Porto
  - Unidade Local de Saude do Alto Minho, EPE, Viana do Castelo
- Romania (11):
  - SC MedLife SA, Gastroenterologie, Bucharest
  - Spitalul Universitar de Urgenta Militar Central Dr. Carol Davila - Sectia Clinica de Gastroenterologie, Bucharest
  - S.C. Centrul Medical Sana S.R.L., Gastroenterologie, Bucharest
  - Delta Health Care/ Ponderas Academic Hospital, Bucharest
  - Spitalul Clinic Colentina, Gastroenterologie, Bucharest
  - MedLife, Gastroenterologie, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti - Sectia Medicina Interna II, Bucharest
  - Gastromedica SRL, Gastroenterologie, Iași
  - Cabinet Particular Policlinic Algomed SRL, Timișoara
  - Centrul Medical Tuculanu, Gastroenterologie, Timișoara
  - S.C. Policlinica Dr. Citu S.R.L.- Gastroenterologie, Timișoara
- Russia (11):
  - State Budgetary Healthcare Institute "Chelyabinsk Regional Clinical Hospital", Chelyabinsk
  - State Budgetary Institution of Health Irkustsk Order "Badge of Honor" Regional Clinical Hospital, Irkutsk
  - State Budgetary Healthcare Institution of Moscow "City Clinical Hospital # 24 of Healthcare Department of Moscow", Moscow
  - State Budgetary Healthcare Institution of Moscow Region "Moscow Regional Clinical Research Institute n.a. M.F. Vladimirskiy", Moscow
  - State Budgetary Healthcare Institution of Nizhny Novgorod Region "Nizhny Novgorod Regional Clinical Hospital n.a. N.A., Nizhny Novgorod
  - State Budgetary Healthcare Institution of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk
  - State Budgetary Institution of Health of Novosibirsk Region "City Clinical Hospital #12", Novosibirsk
  - Saint Petersburg State Budgetary Healthcare Institution "City Polyclinic #38", Saint Petersburg
  - "Scientific Research Centre ECO-safety" LLC, Saint Petersburg
  - "PolyClinic EXPERT" LLC, Saint Petersburg
  - State Healthcare Institution "Regional Clinical Hospital", Saratov
- Serbia (5):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Zvezdara University Medical Center, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (3):
  - Cliniq s. r. o., Gastroenterologicke centrum Ruzinov, Bratislava
  - KM Management, s.r.o., Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Gastro I., s.r.o., Prešov
- South Africa (3):
  - Dr MJ Prins, Cape Town
  - Dr John P Wright, Cape Town
  - Peermed Clinical Trial Centre, Johannesburg
- South Korea (12):
  - Pusan National University Hospital, Busan
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Guri-si
  - Hanyang University Guri Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Division of Gastroenterology, Department of Medicine, Samsung Medical Center, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (13):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Centro Medico Teknon, Barcelona
  - Hospital del Mar, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol
  - Hospital Universitario de Gran Canaria "Dr. Negrin", Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Complejo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital de Galdakao-Usandolo, Usansolo
- Sri Lanka (4):
  - National Hospital of Sri Lanka, Colombo
  - Teaching hospital Karapitiya, Galle
  - Kandy Teaching Hospital, Kandy
  - Colombo North Teaching Hospital, Ragama
- Sweden (2):
  - Danderyds Sjukhus AB, Danderyd
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Gastroenterologische Praxis Balsiger, Seibold und Partner, Bern
  - Universitatsspital Zurich, Zurich
- Taiwan (11):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Chang Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Foundation, Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District
- Ukraine (16):
  - Bukovinian State Medical University, Chernivtsi
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1 st Therapy Department. Danylo Halytsky Lviv National Medical, Chernivtsi
  - State Institution "Institute of Gastroenterology of National Academy of Medical Sciences of Ukraine", Dnipropetrovsk
  - Ivanto-Frankivsk Central City Clinic Hospital, Therapy Department #1. State Higher Education Institution Ivano-Frankivsk National, Ivano-Frankivsk
  - Municipal Health Care Institution "Kharkiv City Clinical Hospital #2 named after prof. O. O. Shalimov", Proctology Department, Kharkiv
  - Municipal Institution of Health Care "Regional Hospital of War Veterans", Therapeutic Department No1, Kharkiv
  - Treatment and Diagnostic Center of Private Enterprise of Private Production Company "Acinus", Kropyvnytskyi
  - Kyiv City Clinical Hospital No. 18, Proctology Department, Kyiv
  - Municipal Non-profit Enterprise "Consultative and Diagnostic Center" of Pechersk District of Kyiv, Therapy Department, Kyiv
  - Municipal Institution "Odesa Regional Clinical Hospital", Regional Gastroenterology Center based on Surgery Department, Odesa
  - Ternopil University Hospital, Regional Center of Gastroenterology with Hepatology, Ternopil
  - Municipal Institution "Uzhgorod District Hospital", Therapy Department, Uzhhorod
  - Vinnytsia Regional Clinical Hospital of War Veterans, Therapy Department #1, Vinnytsia
  - Medical Center LLC "Health Clinic", Vinnytsia
  - M.I. Pyrogov Vinnytsia Regional Clinical Hospital, Gastroenterology Department, Vinnytsia
  - Municipal Institution "Zaporizhzhya Regional Clinical Hospital" of Zaporizhzhya Regional Council, Zaporizhzhya
- United Kingdom (15):
  - Norfolk and Norwich University Hospital NHS Foundation Trust, Norwich, Norfolk
  - Queen Elizabeth Hospital, Birmingham
  - The Pennine Acute Hospitals NHS Trust, Bury
  - Cambridge University Hospital NHS Foundation Trust, Cambridge
  - Royal Derby Hospital, Derby
  - NHS Lothian, Edinburgh
  - Medical Outpatient Department, Exeter
  - Glasgow Clinical Research Facility - Queen Elizabeth University Hospital, Glasgow
  - NHS Greater Glasgow and Clyde, Glasgow
  - Wycombe Hospital, High Wycombe
  - Hull Royal Infirmary, Hull
  - Imperial College Healthcare NHS Trust, St Mary's Hospital, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Southampton National Institute for Health Research, Wellcome Trust Clinical Research Facility, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermeire S, Schreiber S, Rubin DT, D'Haens G, Reinisch W, Watanabe M, Mehta R, Roblin X, Beales I, Gietka P, Hibi T, Hospodarskyy I, Ritter T, Genovese MC, Kwon P, Santermans E, Le Brun FO, Barron R, Masior T, Danese S. Efficacy and safety of filgotinib as induction and maintenance therapy for Crohn's disease (DIVERSITY): a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2025 Feb;10(2):138-153. doi: 10.1016/S2468-1253(24)00272-3. Epub 2024 Dec 2. PMID 39637881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with diagnosis of moderately to severely Active Crohn's disease (CD) were enrolled in the study. Participants who were biologic-naïve or biologic-experienced were enrolled in Cohort A and participants who were biologic-experienced were enrolled in Cohort B, respectively.
Pre-assignment Details: Participants who met protocol eligibility criteria were assigned to the respective Cohort and subsequently randomized in a blinded fashion in a 1:1:1 ratio to 1 of 3 treatments: filgotinib 200 milligram (mg), filgotinib 100 mg and placebo.
Groups:
- Cohort A: Filgotinib 200 mg (Induction Study): Biologic naïve and biologic experienced participants received filgotinib 200 mg with placebo-to-match (PTM) filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
- Placebo to Placebo (Maintenance Study): Participants who received placebo in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
Period: Induction Study (Day 1 to Week 10)
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study) | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 200 mg to Placebo (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) | Filgotinib 100 mg to Placebo (Maintenance Study) | Placebo to Placebo (Maintenance Study)
Started | 223 | 245 | 239 | 204 | 230 | 231 | 0 | 0 | 0 | 0 | 0
Treated | 222 | 245 | 237 | 202 | 228 | 229 | 0 | 0 | 0 | 0 | 0
Completed | 204 | 213 | 212 | 177 | 183 | 192 | 0 | 0 | 0 | 0 | 0
Not Completed | 19 | 32 | 27 | 27 | 47 | 39 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 15 | 14 | 14 | 24 | 31 | 19 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 9 | 6 | 0 | 7 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 4 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 5 | 2 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance with Study Drug | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 1 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Study (Weeks 11 to 58)
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study) | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 200 mg to Placebo (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) | Filgotinib 100 mg to Placebo (Maintenance Study) | Placebo to Placebo (Maintenance Study)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 118 (Not all participants who completed the induction study entered the maintenance study.) | 56 (Not all participants who completed the induction study entered the maintenance study.) | 105 (Not all participants who completed the induction study entered the maintenance study.) | 56 (Not all participants who completed the induction study entered the maintenance study.) | 146 (Not all participants who completed the induction study entered the maintenance study.)
Treated | 0 | 0 | 0 | 0 | 0 | 0 | 118 | 56 | 104 | 55 | 145
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 64 | 21 | 45 | 26 | 74
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 54 | 35 | 60 | 30 | 72
Not completed — Protocol-Specified Disease Worsening | 0 | 0 | 0 | 0 | 0 | 0 | 31 | 32 | 40 | 25 | 43
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 2 | 11 | 2 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2 | 1 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 2 | 0 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The All Randomized Analysis Set included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study) | Total
Number analyzed (Participants) | 223 | 245 | 239 | 204 | 230 | 231 | 1372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 213 | 233 | 229 | 191 | 220 | 227 | 1313
  >=65 years | 10 | 12 | 10 | 13 | 10 | 4 | 59
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 106 | 130 | 115 | 129 | 116 | 706
  Male | 113 | 139 | 109 | 89 | 101 | 115 | 666
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 4 | 2 | 8 | 4 | 27
  Not Hispanic or Latino | 214 | 237 | 232 | 193 | 217 | 220 | 1313
  Unknown or Not Reported | 5 | 3 | 3 | 9 | 5 | 7 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 45 | 52 | 44 | 24 | 25 | 31 | 221
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Black or African American | 3 | 6 | 4 | 6 | 9 | 6 | 34
  White | 166 | 179 | 185 | 158 | 182 | 178 | 1048
  Other | 2 | 3 | 2 | 3 | 0 | 1 | 11
  Unknown or Not Reported | 7 | 5 | 4 | 13 | 12 | 13 | 54
Region of Enrollment [Number; unit: participants]
  Hong Kong | 1 | 0 | 3 | 0 | 0 | 0 | 4
  United States | 22 | 41 | 45 | 51 | 84 | 60 | 303
  Czechia | 2 | 9 | 9 | 1 | 2 | 5 | 28
  Malaysia | 4 | 3 | 0 | 1 | 0 | 0 | 8
  Portugal | 1 | 3 | 1 | 0 | 2 | 2 | 9
  Iceland | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Russia | 7 | 4 | 5 | 3 | 3 | 2 | 24
  Greece | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Austria | 0 | 0 | 0 | 1 | 2 | 0 | 3
  Netherlands | 6 | 3 | 5 | 6 | 7 | 9 | 36
  South Korea | 0 | 2 | 7 | 0 | 4 | 5 | 18
  Sweden | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Ireland | 1 | 1 | 0 | 4 | 0 | 1 | 7
  Poland | 35 | 25 | 34 | 12 | 7 | 12 | 125
  Slovakia | 0 | 3 | 2 | 3 | 3 | 4 | 15
  France | 19 | 15 | 16 | 28 | 21 | 31 | 130
  Serbia | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Croatia | 0 | 1 | 1 | 0 | 1 | 1 | 4
  Romania | 2 | 1 | 3 | 1 | 2 | 0 | 9
  Hungary | 6 | 6 | 2 | 1 | 0 | 1 | 16
  Sri Lanka | 4 | 4 | 3 | 0 | 0 | 1 | 12
  Japan | 8 | 10 | 8 | 12 | 10 | 13 | 61
  Ukraine | 18 | 16 | 20 | 0 | 0 | 0 | 54
  United Kingdom | 5 | 5 | 4 | 6 | 7 | 6 | 33
  Switzerland | 1 | 0 | 6 | 0 | 2 | 4 | 13
  India | 23 | 30 | 20 | 7 | 6 | 5 | 91
  Spain | 5 | 5 | 1 | 5 | 8 | 3 | 27
  New Zealand | 2 | 1 | 3 | 0 | 3 | 2 | 11
  Canada | 9 | 6 | 7 | 7 | 4 | 4 | 37
  Belgium | 6 | 11 | 7 | 15 | 12 | 11 | 62
  Norway | 0 | 1 | 1 | 1 | 1 | 0 | 4
  Taiwan | 4 | 1 | 1 | 1 | 0 | 3 | 10
  Italy | 3 | 8 | 3 | 7 | 6 | 5 | 32
  South Africa | 6 | 1 | 1 | 1 | 0 | 0 | 9
  Georgia | 2 | 1 | 1 | 0 | 0 | 0 | 4
  Israel | 2 | 9 | 2 | 6 | 3 | 7 | 29
  Australia | 11 | 6 | 8 | 4 | 9 | 11 | 49
  Germany | 8 | 10 | 9 | 19 | 18 | 19 | 83
  Singapore | 0 | 0 | 0 | 0 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Induction Study: Percentage of Participants Who Achieved Clinical Remission by Crohn's Disease Activity Index (CDAI) at Week 10
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Clinical remission was defined as a CDAI of < 150 points.
Time Frame: Week 10
Population: The Full Analysis Set (FAS) for each Induction Study (Cohorts A and B) included all randomized participants who took at least 1 dose of study drug in the corresponding Induction Study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A: Filgotinib 200 mg (Induction Study): Biologic naïve and biologic experienced participants received filgotinib 200 mg with PTM filgotinib 100 mg tablet orally once daily, for a period of 10 weeks.
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study)
Number analyzed (Participants) | 222 | 245 | 237 | 202 | 228 | 229
percentage of participants | 32.9 [26.5 to 39.3] | 25.7 [20.0 to 31.4] | 19.8 [14.5 to 25.1] | 26.7 [20.4 to 33.1] | 16.7 [11.6 to 21.7] | 14.8 [10.0 to 19.7]
Statistical Analysis 1: Comparison: Cohort A: Filgotinib 200 mg (Induction Study) vs Cohort A: Placebo (Induction Study); Cochran-Mantel-Haenszel (CMH) test was stratified by concomitant use of oral, systemic corticosteroids (Yes/No) and of immunomodulators (Yes/No) at Day 1, and number of prior exposures to biologic agent (0, >=1); Test type: Superiority; p = 0.0017, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 12.7, 95% CI 2-sided [4.7 to 20.7]
Statistical Analysis 2: Comparison: Cohort A: Filgotinib 100 mg (Induction Study) vs Cohort A: Placebo (Induction Study); CMH test was stratified by concomitant use of oral, systemic corticosteroids (Yes/No) and of immunomodulators (Yes/No) at Day 1, and number of prior exposures to biologic agent (0, >=1); Test type: Superiority; p = 0.1730, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 5.2, 95% CI 2-sided [-2.4 to 12.7]
Statistical Analysis 3: Comparison: Cohort B: Filgotinib 200 mg (Induction Study) vs Cohort B: Placebo (Induction Study); CMH test was stratified by concomitant use of oral, systemic corticosteroids (Yes/No) and of immunomodulators (Yes/No) at Day 1, and number of prior exposures to biologic agent (<=1, >1); Test type: Superiority; p = 0.0023, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 12.0, 95% CI 2-sided [4.1 to 19.9]
Statistical Analysis 4: Comparison: Cohort B: Filgotinib 100 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.6038, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 1.8, 95% CI 2-sided [-5.2 to 8.7]

2. Primary Outcome: Induction Study: Percentage of Participants Who Achieved Endoscopic Response at Week 10
Description: The Simple Endoscopic Score for Crohn's Disease (SES-CD) assessed the degree of inflammation on the basis of 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater severity of disease. Endoscopic response was defined as ≥ 50% reduction from baseline in total SES-CD score.
Time Frame: Week 10
Population: FAS for induction study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study)
Number analyzed (Participants) | 222 | 245 | 237 | 202 | 228 | 229
percentage of participants | 23.9 [18.0 to 29.7] | 20.8 [15.5 to 26.1] | 18.1 [13.0 to 23.3] | 11.9 [7.2 to 16.6] | 13.6 [8.9 to 18.3] | 11.4 [7.0 to 15.7]
Statistical Analysis 1: Comparison: Cohort A: Filgotinib 200 mg (Induction Study) vs Cohort A: Placebo (Induction Study); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.1365, Cochran-Mantel-Haenszel; CMH test stratified by use of corticosteroids (Yes/No), immunomodulators (Yes/No), and prior exposure to biologic agents (0, >=1) at Day 1; Stratified Percentage Difference = 5.5, 95% CI 2-sided [-2.0 to 12.9]
Statistical Analysis 2: Comparison: Cohort A: Filgotinib 100 mg (Induction Study) vs Cohort A: Placebo (Induction Study); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.5103, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 2.4, 95% CI 2-sided [-4.8 to 9.5]
Statistical Analysis 3: Comparison: Cohort B: Filgotinib 200 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.9797, Cochran-Mantel-Haenszel; CMH test stratified by use of corticosteroids (Yes/No), immunomodulators (Yes/No), and prior exposure to biologic agents (<=1, >1) at Day 1; Stratified Percentage Difference = 0.1, 95% CI 2-sided [-6.5 to 6.6]
Statistical Analysis 4: Comparison: Cohort B: Filgotinib 100 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.4264, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 2.4, 95% CI 2-sided [-3.9 to 8.8]

3. Primary Outcome: Maintenance Study: Percentage of Participants Who Achieved Clinical Remission by CDAI at Week 58
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Clinical remission was defined as a CDAI of < 150 points.
Time Frame: Week 58
Population: The FAS for the Maintenance Study included all participants randomized to either the filgotinib 200 mg or filgotinib 100 mg treatment groups in the Induction Studies who were re-randomized in the Maintenance Study and took at least 1 dose of study drug in the Maintenance Study and achieved clinical remission by PRO2 or endoscopic response at Week 10.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study): Participants who received filgotinib 200 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, up to Week 58.
- Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study): Participants who received filgotinib 100 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received filgotinib 100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
- Filgotinib 200 mg - Placebo (Maintenance Study): Participants who received filgotinib 200 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 100 mg and PTM filgotinib 200 mg tablet orally once daily, up to Week 58.
- Filgotinib 100 mg - Placebo (Maintenance Study): Participants who received filgotinib 100 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, up to Week 58.
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 42.9 [33.2 to 52.5] | 23.5 [14.6 to 32.4] | 28.3 [15.2 to 41.4] | 22.6 [10.4 to 34.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); CMH test was stratified by concomitant use of immunomodulators (Yes/No), at Maintenance baseline, and history of exposure to a biologic agent (Yes/No); Test type: Superiority; p = 0.0839, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 13.7, 95% CI 2-sided [-1.0 to 28.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.8288, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 1.5, 95% CI 2-sided [-12.1 to 15.0]

4. Primary Outcome: Maintenance Study: Percentage of Participants Who Achieved Endoscopic Response at Week 58
Description: The SES-CD assessed the degree of inflammation on the basis of 4 components: size of ulcers, ulcerated surface, affected surface, and presence of narrowing. Each of these components was scored on a scale of 0 to 3 (worst). In the SES-CD, each of these 4 components are assessed in the five segments: ileum, right colon, transverse colon, left colon, and rectum. The SES-CD was the sum of the individual scores of each of the components across the five segments. The range of SES-CD scores was 0 - 12 for each segment, and 0 - 60 for the overall SES-CD score, with larger scores indicating greater severity of disease. Endoscopic response was defined as ≥ 50% reduction from baseline in total SES-CD score.
Time Frame: Week 58
Population: The FAS for the Maintenance Study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 30.4 [21.4 to 39.3] | 18.4 [10.2 to 26.5] | 9.4 [0.6 to 18.2] | 13.2 [3.1 to 23.3]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0038, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 20.6, 95% CI 2-sided [8.2 to 33.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.3466, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 5.8, 95% CI 2-sided [-6.6 to 18.3]

5. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved Clinical Remission by PRO2 at Week 10
Description: The PRO2 was a composite score based on 2 components of the CDAI, the number of liquid or soft stools/day for 7 days, stool frequency and abdominal pain (rated on a scale of 0-3) assessed for 7 days. Clinical Remission was defined as the average daily stool score ≤3 points AND average daily abdominal pain score ≤1 point.
Time Frame: Week 10
Population: FAS for induction study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study)
Number analyzed (Participants) | 222 | 245 | 237 | 202 | 228 | 229
percentage of participants | 32.9 [26.5 to 39.3] | 30.6 [24.6 to 36.6] | 25.7 [20.0 to 31.5] | 29.7 [23.2 to 36.3] | 18.9 [13.6 to 24.2] | 17.9 [12.7 to 23.1]
Statistical Analysis 1: Comparison: Cohort A: Filgotinib 200 mg (Induction Study) vs Cohort A: Placebo (Induction Study); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0963, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 6.9, 95% CI 2-sided [-1.4 to 15.2]
Statistical Analysis 2: Comparison: Cohort A: Filgotinib 100 mg (Induction Study) vs Cohort A: Placebo (Induction Study); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3050, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 4.2, 95% CI 2-sided [-3.9 to 12.2]
Statistical Analysis 3: Comparison: Cohort B: Filgotinib 200 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0039, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 11.9, 95% CI 2-sided [3.7 to 20.2]
Statistical Analysis 4: Comparison: Cohort B: Filgotinib 100 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.7556, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 1.1, 95% CI 2-sided [-6.2 to 8.5]

6. Secondary Outcome: Induction Study: Percentage of Participants Who Achieved Clinical Response by CDAI at Week 10
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Clinical response was defined as reduction in CDAI score from Induction baseline by at least 100 points or CDAI score < 150 points.
Time Frame: Week 10
Population: FAS for induction study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study)
Number analyzed (Participants) | 222 | 245 | 237 | 202 | 228 | 229
percentage of participants | 52.3 [45.5 to 59.0] | 46.1 [39.7 to 52.6] | 39.7 [33.2 to 46.1] | 38.6 [31.7 to 45.6] | 35.5 [29.1 to 42.0] | 27.5 [21.5 to 33.5]
Statistical Analysis 1: Comparison: Cohort A: Filgotinib 200 mg (Induction Study) vs Cohort A: Placebo (Induction Study); CMH test was stratified by concomitant use of oral, systemic corticosteroids (Yes/No) and of immunomodulators (Yes/No) at Day 1, and number of prior exposures to biologic agent (0, ≥1); Test type: Superiority; p = 0.0074, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 12.0, 95% CI 2-sided [3.2 to 20.8]
Statistical Analysis 2: Comparison: Cohort A: Filgotinib 100 mg (Induction Study) vs Cohort A: Placebo (Induction Study); [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.2159, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 5.5, 95% CI 2-sided [-3.2 to 14.1]
Statistical Analysis 3: Comparison: Cohort B: Filgotinib 200 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0110, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 11.6, 95% CI 2-sided [2.6 to 20.6]
Statistical Analysis 4: Comparison: Cohort B: Filgotinib 100 mg (Induction Study) vs Cohort B: Placebo (Induction Study); [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0593, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 8.2, 95% CI 2-sided [-0.4 to 16.7]

7. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Clinical Remission by PRO2 at Week 58
Description: as for outcome 5
Time Frame: Week 58
Population: The FAS for the Maintenance Study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 43.8 [34.1 to 53.4] | 29.6 [20.0 to 39.1] | 26.4 [13.6 to 39.2] | 24.5 [12.0 to 37.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0382, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 16.8, 95% CI 2-sided [2.0 to 31.6]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4263, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 5.8, 95% CI 2-sided [-8.5 to 20.0]

8. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Clinical Response by CDAI at Week 58
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Clinical response was defined as reduction in CDAI score from Induction baseline by at least 100 points or CDAI score < 150 points.
Time Frame: Week 58
Population: The FAS for the Maintenance Study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 45.5 [35.9 to 55.2] | 33.7 [23.8 to 43.5] | 34.0 [20.3 to 47.7] | 30.2 [16.9 to 43.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); CMH test was stratified by concomitant use of immunomodulators (Yes/No) at Maintenance baseline, and history of exposure to a biologic agent (Yes/No); Test type: Superiority; p = 0.1827, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 10.9, 95% CI 2-sided [-4.7 to 26.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.5944, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 4.0, 95% CI 2-sided [-11.1 to 19.2]

9. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Sustained Clinical Remission by CDAI at Both Weeks 10 and 58
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The sub scores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  Sustained Clinical Remission by CDAI: CDAI <150 combined at both Week 10 and Week 58.
Time Frame: Weeks 10 and 58
Population: The FAS for the Maintenance Study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 38.4 [28.9 to 47.8] | 19.4 [11.1 to 27.7] | 22.6 [10.4 to 34.9] | 20.8 [8.9 to 32.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0512, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 15.2, 95% CI 2-sided [1.0 to 29.3]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.9801, Cochran-Mantel-Haenszel; Stratified Percentage Difference = -0.2, 95% CI 2-sided [-13.3 to 13.0]

10. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved 6 Month Corticosteroid-Free Remission by CDAI at Week 58
Description: The CDAI system was a composite index of 8 disease activity variables: severity of abdominal pain, general well-being, very soft/liquid stool frequency, extra-intestinal symptoms, need for antidiarrheal drugs, presence of an abdominal mass, body weight and hematocrit. Participants reported information regarding symptoms using a diary. The subscores of abdominal pain (0-3), general well-being (0-4), and number of very soft or liquid stools were then summed over the 7 days prior to each visit. Additionally, the remaining predictors were also noted and weighted to create the total CDAI score which ranged from 0-600 with a higher score indicating a worse outcome.
  6-Month Corticosteroid-Free Clinical remission by CDAI: CDAI <150 with no corticosteroid use for indication of Crohn's disease for at least 6 months prior to Week 58.
Time Frame: Week 58
Population: The FAS for the Maintenance Study with available data was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 50 | 41 | 25 | 25
percentage of participants | 34.0 [19.9 to 48.1] | 4.9 [0.0 to 12.7] | 20.0 [2.3 to 37.7] | 12.0 [0.0 to 26.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); CMH test was stratified by immunomodulators (Yes) at Maintenance baseline, immunomodulators (No) at Maintenance baseline and history of exposure to biologic agent (Yes), and immunomodulators (No) at Maintenance baseline and history of exposure to biologic agent (No); Test type: Superiority; p = 0.1900, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 14.0, 95% CI 2-sided [-5.1 to 33.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.4248, Cochran-Mantel-Haenszel; Stratified Percentage Difference = -5.5, 95% CI 2-sided [-22.6 to 11.6]

11. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved Sustained Clinical Remission by PRO2 at Both Weeks 10 and 58
Description: The PRO2 was a composite score based on 2 components of the CDAI, the number of liquid or soft stools/day for 7 days, stool frequency and abdominal pain (rated on a scale of 0-3) assessed for 7 days.
  Sustained Clinical Remission by PRO2: liquid or very soft stool ≤3 and abdominal pain ≤1 combined at both Week 10 and Week 58.
Time Frame: Weeks 10 and 58
Population: The FAS for the Maintenance Study was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 112 | 98 | 53 | 53
percentage of participants | 41.1 [31.5 to 50.6] | 25.5 [16.4 to 34.7] | 20.8 [8.9 to 32.6] | 24.5 [12.0 to 37.1]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); CMH test was stratified by concomitant use immunomodulators (Yes/No), at Maintenance baseline, and history of exposure to a biologic agent (Yes/No); Test type: Superiority; p = 0.0122, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 19.9, 95% CI 2-sided [5.7 to 34.0]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.7708, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 2.0, 95% CI 2-sided [-12.0 to 16.1]

12. Secondary Outcome: Maintenance Study: Percentage of Participants Who Achieved 6 Month Corticosteroid-Free Remission by PRO2 at Week 58
Description: The PRO2 was a composite score based on 2 components of the CDAI, the number of liquid or soft stools/day for 7 days, stool frequency and abdominal pain (rated on a scale of 0-3) assessed for 7 days.
  6-month Corticosteroid-Free Clinical Remission by PRO2: liquid or very soft stool ≤3 and abdominal pain ≤1 with no corticosteroid use for at least 6 months prior to Week 58.
Time Frame: Week 58
Population: The FAS for the Maintenance Study with available data was analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) | Filgotinib 200 mg - Placebo (Maintenance Study) | Filgotinib 100 mg - Placebo (Maintenance Study)
Number analyzed (Participants) | 50 | 41 | 25 | 25
percentage of participants | 32.0 [18.1 to 45.9] | 7.3 [0.0 to 16.5] | 20.0 [2.3 to 37.7] | 12.0 [0.0 to 26.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg - Filgotinib 200 mg (Maintenance Study) vs Filgotinib 200 mg - Placebo (Maintenance Study); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.2631, Cochran-Mantel-Haenszel; Stratified Percentage Difference = 12.0, 95% CI 2-sided [-8.3 to 32.3]
Statistical Analysis 2: Comparison: Filgotinib 100 mg - Filgotinib 100 mg (Maintenance Study) vs Filgotinib 100 mg - Placebo (Maintenance Study); [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.6444, Cochran-Mantel-Haenszel; Stratified Percentage Difference = -3.4, 95% CI 2-sided [-20.9 to 14.0]

13. Secondary Outcome: Induction Study:Pharmacokinetic Plasma Concentrations of Filgotinib at Week 4
Description: Plasma concentrations of filgotinib [nanogram/milliliters (ng/mL)].
Time Frame: Week 4: 0.5, 1, 2, and 3 hours (hrs) post dose
Population: Pharmacokinetic (PK) Analysis Set (included all randomized participants who took at least 1 dose of filgotinib and had at least 1 non-missing concentration value for filgotinib and/or its metabolite GS-829845 reported by the PK laboratory) for Induction study was analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study)
Number analyzed (Participants) | 177 | 181 | 141 | 168
ng/mL | 1170 (1270) | 611 (634) | 1140 (1070) | 604 (634)

14. Secondary Outcome: Induction Study: Pharmacokinetic Plasma Concentrations of Filgotinib at Week 10
Description: Plasma concentrations of filgotinib (ng/mL).
Time Frame: Week 10: Predose
Population: PK Analysis Set for Induction study was analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study)
Number analyzed (Participants) | 183 | 180 | 136 | 135
ng/mL | 46.8 (180) | 21.3 (79.5) | 47.9 (215) | 40.8 (139)

15. Secondary Outcome: Maintenance Study: Pharmacokinetic Plasma Concentrations of Filgotinib at Week 26
Description: Plasma concentrations of filgotinib (ng/mL).
Time Frame: Week 26: At any timepoint
Population: PK Analysis Set for Maintenance study was analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study)
Number analyzed (Participants) | 77 | 63
ng/mL | 284 (623) | 58.5 (150)

16. Secondary Outcome: Maintenance Study: Pharmacokinetic Plasma Concentrations of Filgotinib at Week 58
Description: Plasma concentrations of filgotinib (ng/mL).
Time Frame: Week 58: Pre-dose
Population: PK Analysis Set for Maintenance study was analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study)
Number analyzed (Participants) | 34 | 27
ng/mL | 75.8 (238) | 16.9 (55.5)

17. Secondary Outcome: Induction Study: Pharmacokinetic Plasma Concentrations of Filgotinib's Metabolite GS-829845 at Week 4
Description: Plasma concentrations of GS-829845 (ng/mL).
Time Frame: Week 4: 0.5, 1, 2, and 3 hrs post dose
Population: PK Analysis Set for Induction study was analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study)
Number analyzed (Participants) | 177 | 181 | 141 | 168
ng/mL | 3100 (1530) | 1800 (936) | 3140 (1450) | 1870 (776)

18. Secondary Outcome: Induction Study: Pharmacokinetic Plasma Concentrations of Filgotinib's Metabolite GS-829845 at Week 10
Description: Plasma concentrations of GS-829845 (ng/mL).
Time Frame: Week 10: Predose
Population: PK Analysis Set for Induction study was analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study)
Number analyzed (Participants) | 183 | 180 | 136 | 135
ng/mL | 2550 (1390) | 1290 (801) | 2640 (1470) | 1480 (917)

19. Secondary Outcome: Maintenance Study: Pharmacokinetic Plasma Concentrations of Filgotinib's Metabolite GS-829845 at Week 26
Description: Plasma concentrations of GS-829845 (ng/mL).
Time Frame: Week 26: At any timepoint
Population: PK Analysis Set for Maintenance study was analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study)
Number analyzed (Participants) | 77 | 63
ng/mL | 3090 (1500) | 1460 (814)

20. Secondary Outcome: Maintenance Study: Pharmacokinetic Plasma Concentrations of Filgotinib's Metabolite GS-829845 at Week 58
Description: Plasma concentrations of GS-829845 (ng/mL).
Time Frame: Week 58: Pre-dose
Population: PK Analysis Set for Maintenance study was analyzed
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study)
Number analyzed (Participants) | 34 | 27
ng/mL | 2430 (1430) | 1220 (551)

ADVERSE EVENTS:
Time Frame: From first dose up to Week 62
Description: Safety Analysis Set
Groups:
- Filgotinib 200 mg to Placebo (Maintenance Study): Participants who received filgotinib 200 mg in induction study and who achieved either clinical remission by PRO2 or endoscopic response at Week 10 were re-randomized to the maintenance study and received PTM filgotinib 200 mg and PTM filgotinib 100 mg tablet orally once daily, up to Week 58.
Arm/Group | Cohort A: Filgotinib 200 mg (Induction Study) | Cohort A: Filgotinib 100 mg (Induction Study) | Cohort A: Placebo (Induction Study) | Cohort B: Filgotinib 200 mg (Induction Study) | Cohort B: Filgotinib 100 mg (Induction Study) | Cohort B: Placebo (Induction Study) | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) | Filgotinib 200 mg to Placebo (Maintenance Study) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) | Filgotinib 100 mg to Placebo (Maintenance Study) | Placebo to Placebo (Maintenance Study)
All-Cause Mortality (participants affected / at risk) | 0/222 | 0/245 | 0/237 | 0/202 | 0/228 | 0/229 | 0/118 | 0/56 | 0/104 | 0/55 | 0/145
Serious Adverse Events (participants affected / at risk) | 18/222 | 16/245 | 15/237 | 19/202 | 36/228 | 26/229 | 13/118 | 5/56 | 14/104 | 3/55 | 14/145
Other Adverse Events (participants affected / at risk) | 87/222 | 90/245 | 90/237 | 106/202 | 107/228 | 109/229 | 59/118 | 28/56 | 59/104 | 25/55 | 77/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Filgotinib 200 mg (Induction Study) (N=222) | Cohort A: Filgotinib 100 mg (Induction Study) (N=245) | Cohort A: Placebo (Induction Study) (N=237) | Cohort B: Filgotinib 200 mg (Induction Study) (N=202) | Cohort B: Filgotinib 100 mg (Induction Study) (N=228) | Cohort B: Placebo (Induction Study) (N=229) | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) (N=118) | Filgotinib 200 mg to Placebo (Maintenance Study) (N=56) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) (N=104) | Filgotinib 100 mg to Placebo (Maintenance Study) (N=55) | Placebo to Placebo (Maintenance Study) (N=145)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza A virus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central serous chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal scar (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 7 (7) | 9 (9) | 7 (8) | 9 (9) | 10 (10) | 10 (10) | 3 (3) | 2 (2) | 7 (7) | 1 (1) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Megacolon (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis enteropathic (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral spondyloarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Primary adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Peritoneal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Filgotinib 200 mg (Induction Study) (N=222) | Cohort A: Filgotinib 100 mg (Induction Study) (N=245) | Cohort A: Placebo (Induction Study) (N=237) | Cohort B: Filgotinib 200 mg (Induction Study) (N=202) | Cohort B: Filgotinib 100 mg (Induction Study) (N=228) | Cohort B: Placebo (Induction Study) (N=229) | Filgotinib 200 mg to Filgotinib 200 mg (Maintenance Study) (N=118) | Filgotinib 200 mg to Placebo (Maintenance Study) (N=56) | Filgotinib 100 mg to Filgotinib 100 mg (Maintenance Study) (N=104) | Filgotinib 100 mg to Placebo (Maintenance Study) (N=55) | Placebo to Placebo (Maintenance Study) (N=145)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 8 (8) | 7 (7) | 6 (7) | 8 (8) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1) | 4 (5)
Weight decreased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 4 (5) | 5 (6) | 4 (4) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7) | 4 (4) | 4 (4) | 7 (7) | 1 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 16 (17) | 12 (12) | 17 (19) | 14 (15) | 15 (18) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 10 (13)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 4 (5) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (3) | 3 (3) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 3 (4) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 16 (16) | 6 (6) | 8 (8) | 10 (14) | 8 (12) | 15 (15) | 8 (8) | 6 (9) | 9 (9) | 3 (3) | 9 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 4 (4) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 5 (5) | 15 (15) | 16 (16) | 8 (8) | 14 (16) | 18 (18) | 15 (16) | 10 (10) | 22 (24) | 15 (15) | 26 (26)
Aphthous ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (4) | 1 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2 (2) | 4 (4) | 7 (7) | 5 (5) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 10 (10) | 11 (11) | 20 (21) | 10 (12) | 18 (19) | 6 (6) | 3 (4) | 3 (3) | 2 (3) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 6 (6) | 6 (6) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 11 (12) | 6 (7) | 7 (10) | 14 (14) | 9 (15) | 3 (3) | 2 (4) | 10 (12) | 4 (5) | 10 (11)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (7) | 7 (8) | 5 (11) | 6 (7) | 9 (9) | 5 (5) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 2 (2) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Bronchitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 4 (4) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 4 (4)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 7 (8) | 6 (6) | 8 (9) | 9 (9) | 9 (11) | 17 (18) | 6 (11) | 4 (4) | 6 (6) | 2 (2) | 9 (9)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 5 (5) | 4 (4) | 10 (11) | 9 (9) | 5 (6) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 5 (6) | 10 (11) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1)
Seborrheic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 3 (3) | 5 (5) | 4 (4) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Asthenia (General disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 8 (9) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (7) | 5 (5) | 4 (4) | 3 (3) | 6 (6) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3)
Pyrexia (General disorders) | 10 (11) | 10 (10) | 6 (7) | 11 (17) | 8 (8) | 10 (12) | 6 (6) | 4 (4) | 3 (4) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT02914561/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02914561/SAP_001.pdf